CLINICAL TRIAL: NCT01587040
Title: International, Multicenter, Open-label, Treatment-extension Study for Subjects Who Completed a Phase 1 or Phase 2 Parental Study to Continue Receiving Treatment With SAR245408 or SAR245409 as a Monotherapy or as a Combination Regimen
Brief Title: Open Label Treatment Extension Study With SAR245408 or SAR245409 as a Monotherapy or as a Combination Regimen
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TED12414; 2011-006140-78 (EudraCT Number); U1111-1124-1403 (Other: UTN)
Record Dates: First submitted 2012-04-25; First posted 2012-04-27 (Estimated); Results first posted 2019-06-11 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Neoplasm Malignant
MeSH Terms: conditions — Neoplasms | interventions — XL147; XL765

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- SAR245408: Monotherapy (Experimental): Participants received SAR245408 400 milligrams (mg) once daily or at the established dose as monotherapy in the parental study until disease progression, unacceptable toxicity, withdrawal of consent, or until commercial supplies of SAR245408 were available (up to 1959 days).
  Interventions: Drug: SAR245408
- SAR245408: Combination Regimen (Experimental): Participants received SAR245408 400 mg once daily or at the established dose as combination regimen in the parental study until disease progression, unacceptable toxicity, withdrawal of consent, or until commercial supplies of SAR245408 were available (up to 1959 days). Commercially available drugs were used as combination medications with SAR245408 (depending on the parental study, the following drugs were used in combination with SAR245408: paclitaxel and carboplatin, letrozole, trastuzumab, paclitaxel and trastuzumab).
  Interventions: Drug: SAR245408
- SAR245409: Monotherapy (Experimental): Participants received SAR245409 50 mg twice daily or at the established dose as monotherapy in the parental study until disease progression, unacceptable toxicity, withdrawal of consent, or until commercial supplies of SAR245409 were available (up to 1917 days).
  Interventions: Drug: SAR245409
- SAR245409: Combination Regimen (Experimental): Participants received SAR245409 50 mg twice daily or at the established dose as combination regimen in the parental study until disease progression, unacceptable toxicity, withdrawal of consent, or until commercial supplies of SAR245409 were available (up to 1917 days). Commercially available drugs were used as combination medications with SAR245409 (depending on the parental study, the following drugs were used in combination with SAR245409: letrozole, temozolomide, rituximab, bendamustine and rituximab).
  Interventions: Drug: SAR245409

INTERVENTIONS:
Drug: SAR245408 — Pharmaceutical form: capsule or tablet Route of administration: oral
  Arms: SAR245408: Combination Regimen; SAR245408: Monotherapy
Drug: SAR245409 — Pharmaceutical form: capsule or tablet Route of administration: oral
  Arms: SAR245409: Combination Regimen; SAR245409: Monotherapy

SUMMARY:
Primary Objective:

The purpose of this study was to determine the long term safety and tolerability of SAR245408 and SAR245409 as a monotherapy or as part of a combination regimen in participants who were benefiting from treatment.

DETAILED DESCRIPTION:
The duration of the study for an individual participant included:

1. Baseline assessments: within 7 days prior to the first dose of investigational medicinal product (IMP).
2. Study treatment period(s):

   Participants started study treatment at the beginning of the initiation or extension periods based on the length of prior therapy with SAR245408 or SAR245409
   * if <2 cycles, started with initiation period; Participant must have had completed all the visits in the initiation period before moving to the extension period.
   * if >=2 cycles, started with extension period; duration of extension period was unlimited.
   * Participants who took a SAR245408 or SAR245409 daily dose higher than their established dose of SAR245408 or SAR245409, respectively, in the parental study entered the study on Day 1 of the initiation period.
   * Participants who had dose interrupted in the parental study but fulfilled parental protocol criteria to restart IMP treatment entered the treatment-extension study on Day 1 of the initiation period.
   * Participants who fulfilled the parental study criteria for IMP treatment continuation but had ongoing Grade 2 adverse events (AEs) entered the treatment-extension study on Day 1 of the initiation period.

   Participants continued to receive study treatment until disease progression, unacceptable toxicity, withdrawal of consent, or until commercial supplies of SAR245408 or SAR245409 were available to them outside of the clinical trial.
3. Follow-up assessments: 23 to 37 days after the last dose of IMP.

ELIGIBILITY:
Inclusion criteria :

I 01. Males or females enrolled in Phase 1 or Phase 2 studies of SAR245408 or SAR245409 as monotherapy or in combination with other regimens who had completed data collection for the primary endpoint(s) of the parental study or who were being treated beyond the parental study cut-off and meet all the criteria to continue to be treated per the parental protocol.

I 02. All sexually active participants (male and female) must agreed to continue to use accepted methods of barrier contraception (i.e., condoms) during the course of the study and for 3 months after discontinuation of study treatment. For women of childbearing potential and for men who could father a child, a second method of contraception in addition to a barrier method is recommended. Hormonal contraception should be avoided in participants taking SAR245408 due to possible drug-drug interaction.

I 03. Female participants of childbearing potential must had a negative pregnancy test at baseline. Females of childbearing potential were defined as sexually mature women without prior hysterectomy or who had any evidence of menses in the past 12 months. However, women who had been amenorrheic for 12 or more months were still considered to be of childbearing potential if the amenorrhea was possibly due to other causes, including prior chemotherapy, anti-estrogens, or ovarian suppression.

Exclusion criteria:

E 01. The participant discontinued the parental study due to toxicity. E 02. Ongoing Grade 3 or higher Adverse Event (AE). E 03. Ongoing Serious Adverse Event (SAE). E 04. Participants with ongoing dose interruption for any reason unless the participant fulfilled the criteria in the parental protocol for restarting IMP. In such case participant started the treatment-extension study on Day 1 of the initiation period.

E 05. The participant had any of the following laboratory values ≥ Common Terminology of Adverse Events (CTCAE) Grade 3

* Absolute neutrophil count (ANC),
* Platelet count,
* Hemoglobin,
* Bilirubin,
* Serum creatinine or calculated creatinine clearance,
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST),
* Fasting plasma glucose (FPG),
* Prothrombin time/international normalized ratio (PT/INR) and activated partial thromboplastin time (aPTT).

E 06. The participant had a baseline corrected QT interval (QTc) >481 millisecond (msec) or if a participant has had a QTc interval increase of ≥ 60 msec from parental protocol baseline to an absolute value of > 470 msec.

E 07. The participant had a known allergy or hypersensitivity to components of the study treatment formulation(s).

E 08. The participant was pregnant or breastfeeding.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-07-20 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (21):
- United States (16):
  - Investigational Site Number 840010, Birmingham, Alabama
  - Investigational Site Number 840009, Los Angeles, California
  - Investigational Site Number 840008, Los Angeles, California
  - Investigational Site Number 840022, Denver, Colorado
  - Investigational Site Number 840104, Fort Myers, Florida
  - Investigational Site Number 840006, Augusta, Georgia
  - Investigational Site Number 840004, Boston, Massachusetts
  - Investigational Site Number 840021, St Louis, Missouri
  - Investigational Site Number 840002, New Brunswick, New Jersey
  - Investigational Site Number 840020, Canton, Ohio
  - Investigational Site Number 840015, Columbus, Ohio
  - Investigational Site Number 840017, Philadelphia, Pennsylvania
  - Investigational Site Number 840007, Nashville, Tennessee
  - Investigational Site Number 840003, Dallas, Texas
  - Investigational Site Number 840005, San Antonio, Texas
  - Investigational Site Number 840018, Morgantown, West Virginia
- Investigational Site Number 056001, Leuven, Belgium
- France (3):
  - Investigational Site Number 250004, Montpellier
  - Investigational Site Number 250003, Pierre-Bénite
  - Investigational Site Number 250005, Rouen
- Investigational Site Number 724001, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 21 centers in 4 countries between 20 July 2012 and 23 May 2018. Participants who received SAR245408/SAR245409 (IMP) in parental studies (TED12471 [NCT01596270], ARD11437 [NCT01082068], TED12863 [NCT01943838]) were included in study. A total of 67 participants were screened and 61 participants were enrolled in this study.
Pre-assignment Details: Participants who received IMP for <2 cycles in parental study, and participants who took a daily dose of IMP higher than their established dose entered treatment-extension study on Day 1 of initiation period; participants who received IMP >=2 cycles in parental study entered treatment-extension study on Day 1 of extension period.
Period: Overall Study
Arm/Group | SAR245408: Monotherapy | SAR245408: Combination Regimen | SAR245409: Monotherapy | SAR245409: Combination Regimen
Started | 17 | 3 | 37 | 4
Completed | 0 | 0 | 0 | 0
Not Completed | 17 | 3 | 37 | 4
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Adverse Event | 0 | 1 | 10 | 0
Not completed — Disease progression | 12 | 1 | 15 | 3
Not completed — Other than specified | 5 | 1 | 11 | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed on safety population that included all participants who took at least 1 dose of study drug during the study.
Groups:
- SAR245408: Monotherapy: Participants received SAR245408 400 mg once daily or at the established dose as monotherapy in the parental study until disease progression, unacceptable toxicity, withdrawal of consent, or until commercial supplies of SAR245408 were available (up to 1959 days).
- Total: Total of all reporting groups
Arm/Group | SAR245408: Monotherapy | SAR245408: Combination Regimen | SAR245409: Monotherapy | SAR245409: Combination Regimen | Total
Number analyzed (Participants) | 17 | 3 | 37 | 4 | 61
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.6 (13.1) | 53.7 (2.1) | 62.4 (12.0) | 50.0 (15.8) | 61.0 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 3 | 16 | 0 | 31
  Male | 5 | 0 | 21 | 4 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 0 | 3
  Not Hispanic or Latino | 17 | 2 | 35 | 4 | 58
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 0 | 5 | 0 | 8
  White | 14 | 2 | 31 | 4 | 51
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs)
Description: Any untoward medical occurrence in a participant who received IMP was considered an AE without regard to possibility of causal relationship with this treatment. Serious adverse event (SAE): any untoward medical occurrence that resulted in any of the following outcomes: death, life-threatening, required initial/prolonged in-patient hospitalization, persistent/significant disability/incapacity, congenital anomaly/birth defect/considered as medically important event. TEAEs: AEs that developed/worsened/became serious during on-treatment period (time from IMP until 30 days after last dose of any IMP). Any TEAE included participants with both SAE & non-SAEs. TEAE included participants with any treatment-emergent SAE (TESAE). TEAEs that led to death, dose reduction and/or delay, discontinuation & AEs related to treatment were reported. Grades (3=severe, 4=life-threatening/disabling) represents severity of AEs.
Time Frame: From Baseline up to 30 days after the last dose (maximum exposure: 1959 days)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | SAR245408: Monotherapy | SAR245408: Combination Regimen | SAR245409: Monotherapy | SAR245409: Combination Regimen
Number analyzed (Participants) | 17 | 3 | 37 | 4
Participants
  Any TEAE | 16 | 3 | 35 | 3
  Any Grade 3-4 TEAEs | 12 | 2 | 19 | 1
  Any related TEAEs | 12 | 3 | 23 | 2
  Any Grade 3-4 related TEAE | 3 | 0 | 11 | 0
  Any Serious TEAE | 9 | 1 | 10 | 0
  Any Grade 3-4 TESAE | 9 | 1 | 9 | 0
  Any related TESAE | 2 | 0 | 1 | 0
  Any Grade 3-4 related TESAE | 2 | 0 | 0 | 0
  Any TEAE leading to death | 0 | 0 | 3 | 0
  Any TEAE leading to permanent discontinuation | 1 | 1 | 8 | 0
  Any TEAE leading to dose reduction | 3 | 1 | 9 | 1
  Any TEAE leading to dose delay or interruption | 6 | 2 | 16 | 0

2. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Hematological Parameters
Description: Hematological parameters assessed were anemia, neutropenia and thrombocytopenia. Parameters were assessed as per the National Cancer Institute Common Terminology Criteria for Adverse Experience version 4.03 (NCI-CTCAE v 4.03), where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From Baseline up to 30 days after the last dose (maximum exposure: 1959 days)
Population: Analysis was performed on safety population. Here, "Overall number of participants analyzed" = participants with available data for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR245408: Monotherapy | SAR245408: Combination Regimen | SAR245409: Monotherapy | SAR245409: Combination Regimen
Number analyzed (Participants) | 16 | 3 | 36 | 4
Participants
  Anemia: All grades | 13 | 1 | 23 | 1
  Anemia: Grade 1 | 6 | 1 | 18 | 1
  Anemia: Grade 2 | 3 | 0 | 2 | 0
  Anemia: Grade 3 | 4 | 0 | 3 | 0
  Anemia: Grade 4 | 0 | 0 | 0 | 0
  Neutropenia: All grades | 7 | 0 | 10 | 1
  Neutropenia: Grade 1 | 2 | 0 | 5 | 1
  Neutropenia: Grade 2 | 2 | 0 | 1 | 0
  Neutropenia: Grade 3 | 2 | 0 | 2 | 0
  Neutropenia: Grade 4 | 1 | 0 | 2 | 0
  Thrombocytopenia: All grades | 8 | 0 | 20 | 3
  Thrombocytopenia: Grade 1 | 5 | 0 | 17 | 3
  Thrombocytopenia: Grade 2 | 0 | 0 | 2 | 0
  Thrombocytopenia: Grade 3 | 0 | 0 | 0 | 0
  Thrombocytopenia: Grade 4 | 3 | 0 | 1 | 0

3. Primary Outcome: Number of Participants With Potentially Clinically Significant Laboratory Abnormalities: Biochemical Parameters
Description: Biochemical parameters assessed were hyperglycemia, aspartate aminotransferase (ASAT) increased, alanine aminotransferase (ALAT) increased, hyperbilirubinemia, hypocalcemia, creatinine increased. Parameters were assessed as per the NCI-CTCAE v 4.03, where Grade 1 = Mild; Grade 2 = Moderate; Grade 3 = Severe; Grade 4 = Potentially Life Threatening. Grade refers to the severity of the AEs.
Time Frame: From Baseline up to 30 days after the last dose (maximum exposure: 1959 days)
Population: Analysis was performed on safety population. Here, "number analyzed"= participants with available data for specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | SAR245408: Monotherapy | SAR245408: Combination Regimen | SAR245409: Monotherapy | SAR245409: Combination Regimen
Number analyzed (Participants) | 17 | 3 | 37 | 4
Participants
  Hyperglycemia: All Grades: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hyperglycemia: All Grades | 13 | 3 | 25 | 1
  Hyperglycemia: Grade 1: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hyperglycemia: Grade 1 | 11 | 2 | 19 | 1
  Hyperglycemia: Grade 2: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hyperglycemia: Grade 2 | 0 | 1 | 6 | 0
  Hyperglycemia: Grade 3: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hyperglycemia: Grade 3 | 2 | 0 | 0 | 0
  Hyperglycemia: Grade 4: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hyperglycemia: Grade 4 | 0 | 0 | 0 | 0
  ASAT Increased: All Grades: number analyzed (Participants) | 16 | 3 | 36 | 4
  ASAT Increased: All Grades | 7 | 2 | 20 | 1
  ASAT Increased: Grade 1: number analyzed (Participants) | 16 | 3 | 36 | 4
  ASAT Increased: Grade 1 | 6 | 1 | 16 | 1
  ASAT Increased: Grade 2: number analyzed (Participants) | 16 | 3 | 36 | 4
  ASAT Increased: Grade 2 | 1 | 1 | 2 | 0
  ASAT Increased: Grade 3: number analyzed (Participants) | 16 | 3 | 36 | 4
  ASAT Increased: Grade 3 | 0 | 0 | 2 | 0
  ASAT Increased: Grade 4: number analyzed (Participants) | 16 | 3 | 36 | 4
  ASAT Increased: Grade 4 | 0 | 0 | 0 | 0
  ALAT Increased: All Grades: number analyzed (Participants) | 16 | 3 | 36 | 4
  ALAT Increased: All Grades | 5 | 2 | 12 | 0
  ALAT Increased: Grade 1: number analyzed (Participants) | 16 | 3 | 36 | 4
  ALAT Increased: Grade 1 | 4 | 1 | 8 | 0
  ALAT Increased: Grade 2: number analyzed (Participants) | 16 | 3 | 36 | 4
  ALAT Increased: Grade 2 | 1 | 1 | 1 | 0
  ALAT Increased: Grade 3: number analyzed (Participants) | 16 | 3 | 36 | 4
  ALAT Increased: Grade 3 | 0 | 0 | 3 | 0
  ALAT Increased: Grade 4: number analyzed (Participants) | 16 | 3 | 36 | 4
  ALAT Increased: Grade 4 | 0 | 0 | 0 | 0
  Blood Bilirubin Increased:All Grades: number analyzed (Participants) | 15 | 3 | 36 | 4
  Blood Bilirubin Increased:All Grades | 1 | 0 | 9 | 1
  Blood Bilirubin Increased:Grade 1: number analyzed (Participants) | 15 | 3 | 36 | 4
  Blood Bilirubin Increased:Grade 1 | 0 | 0 | 4 | 1
  Blood Bilirubin Increased:Grade 2: number analyzed (Participants) | 15 | 3 | 36 | 4
  Blood Bilirubin Increased:Grade 2 | 0 | 0 | 3 | 0
  Blood Bilirubin Increased:Grade 3: number analyzed (Participants) | 15 | 3 | 36 | 4
  Blood Bilirubin Increased:Grade 3 | 1 | 0 | 2 | 0
  Blood Bilirubin Increased:Grade 4: number analyzed (Participants) | 15 | 3 | 36 | 4
  Blood Bilirubin Increased:Grade 4 | 0 | 0 | 0 | 0
  Hypocalcemia: All Grades: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hypocalcemia: All Grades | 6 | 1 | 7 | 0
  Hypocalcemia: Grade 1: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hypocalcemia: Grade 1 | 4 | 1 | 5 | 0
  Hypocalcemia: Grade 2: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hypocalcemia: Grade 2 | 1 | 0 | 0 | 0
  Hypocalcemia: Grade 3: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hypocalcemia: Grade 3 | 1 | 0 | 2 | 0
  Hypocalcemia: Grade 4: number analyzed (Participants) | 16 | 3 | 36 | 4
  Hypocalcemia: Grade 4 | 0 | 0 | 0 | 0
  Creatinine increased: All Grades: number analyzed (Participants) | 16 | 3 | 36 | 4
  Creatinine increased: All Grades | 5 | 1 | 15 | 0
  Creatinine increased: Grade 1: number analyzed (Participants) | 16 | 3 | 36 | 4
  Creatinine increased: Grade 1 | 3 | 1 | 8 | 0
  Creatinine increased: Grade 2: number analyzed (Participants) | 16 | 3 | 36 | 4
  Creatinine increased: Grade 2 | 1 | 0 | 4 | 0
  Creatinine increased: Grade 3: number analyzed (Participants) | 16 | 3 | 36 | 4
  Creatinine increased: Grade 3 | 0 | 0 | 2 | 0
  Creatinine increased: Grade 4: number analyzed (Participants) | 16 | 3 | 36 | 4
  Creatinine increased: Grade 4 | 1 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: All AEs were collected from the date of signing the consent up to 30 days after the last dose (maximum of 1959 days) regardless of seriousness or relationship to investigational product.
Description: Reported AEs and deaths are TEAEs that is AEs and deaths that developed/worsened during the 'on treatment period' (time from the first dose of any study drug up to 30 days after the last dose of any study drug). Analysis was performed on safety population.
Arm/Group | SAR245408: Monotherapy | SAR245408: Combination Regimen | SAR245409: Monotherapy | SAR245409: Combination Regimen
All-Cause Mortality (participants affected / at risk) | 1/17 | 0/3 | 3/37 | 0/4
Serious Adverse Events (participants affected / at risk) | 9/17 | 1/3 | 10/37 | 0/4
Other Adverse Events (participants affected / at risk) | 15/17 | 3/3 | 34/37 | 3/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR245408: Monotherapy (N=17) | SAR245408: Combination Regimen (N=3) | SAR245409: Monotherapy (N=37) | SAR245409: Combination Regimen (N=4)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina Unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Upper Gastrointestinal Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Disease Progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Systemic Inflammatory Response Syndrome (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholangitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Catheter Site Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral Discitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Staphylococcal Skin Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Femur Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Troponin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Lysis Syndrome (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Myeloid Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haemorrhage Intracranial (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal Colic (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Respiratory Distress (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAR245408: Monotherapy (N=17) | SAR245408: Combination Regimen (N=3) | SAR245409: Monotherapy (N=37) | SAR245409: Combination Regimen (N=4)
Anaemia (Blood and lymphatic system disorders) | 3 (4) | 1 (1) | 2 (2) | 0 (0)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coronary Artery Disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus Bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Ventricular Extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ventricular Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen Impaction (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deafness Unilateral (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ear Discomfort (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperacusis (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Corneal Scar (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retinal Vein Occlusion (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Visual Impairment (Eye disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Vitreous Floaters (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Distension (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal Tenderness (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal Wall Haematoma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anal Incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chapped Lips (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 4 (4) | 1 (1) | 7 (7) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 7 (8) | 2 (2) | 14 (14) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Faeces Discoloured (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 3 (4) | 0 (0) | 2 (2) | 0 (0)
Hypoaesthesia Oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 2 (2) | 10 (10) | 0 (0)
Pancreatic Failure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peptic Ulcer Haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Salivary Gland Enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Short-Bowel Syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (2) | 7 (7) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Catheter Site Discharge (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Face Oedema (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Facial Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 8 (9) | 1 (1) | 8 (8) | 0 (0)
Gait Disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
General Physical Health Deterioration (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Localised Oedema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mucosal Inflammation (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Non-Cardiac Chest Pain (General disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Oedema Peripheral (General disorders) | 3 (3) | 1 (1) | 4 (4) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Performance Status Decreased (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Peripheral Swelling (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 4 (4) | 1 (1) | 6 (6) | 0 (0)
Suprapubic Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contrast Media Allergy (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abscess Limb (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chronic Sinusitis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Gastrointestinal Viral Infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatitis C (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Lower Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Onychomycosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral Candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Postoperative Wound Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory Tract Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 5 (5) | 1 (1)
Skin Infection (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Tooth Abscess (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 3 (3) | 0 (0) | 8 (8) | 1 (1)
Urinary Tract Infection (Infections and infestations) | 2 (2) | 1 (1) | 6 (6) | 0 (0)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Accidental Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Incision Site Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Limb Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Abrasion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Wound Dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Alanine Aminotransferase Increased (Investigations) | 0 (0) | 2 (2) | 4 (5) | 0 (0)
Amylase Increased (Investigations) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 2 (2) | 3 (3) | 0 (0)
Bilirubin Conjugated Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Alkaline Phosphatase Increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Blood Bilirubin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Cholesterol Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine Increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blood Lactate Dehydrogenase Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Phosphorus Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood Urea Increased (Investigations) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Body Temperature Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath Sounds Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Breath Sounds Absent (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac Murmur (Investigations) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Chest X-Ray Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram Qt Prolonged (Investigations) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Heart Rate Irregular (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
International Normalised Ratio Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lipase Increased (Investigations) | 2 (2) | 0 (0) | 8 (8) | 0 (0)
Neutrophil Count Decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nuclear Magnetic Resonance Imaging Brain Abnormal (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Procalcitonin Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Protein Urine Present (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Prothrombin Time Prolonged (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red Blood Cell Count Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Red Blood Cells Urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine Analysis Abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urine Protein/Creatinine Ratio Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vitamin B12 Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D Decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
Weight Increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 1 (2) | 1 (1) | 1 (1) | 0 (0)
White Blood Cell Count Increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
White Blood Cells Urine (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
White Blood Cells Urine Positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 5 (5) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Metabolic Acidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vitamin D Deficiency (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1) | 4 (4) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0)
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Pain In Jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pathological Fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pubic Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scoliosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Squamous Cell Carcinoma Of Skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tumour Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cognitive Disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 3 (3) | 0 (0) | 2 (2) | 1 (1)
Dizziness Postural (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 6 (6) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Memory Impairment (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neuropathy Peripheral (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Partial Seizures (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tremor (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Visual Field Defect (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombosis In Device (Product Issues) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0) | 4 (4) | 0 (0)
Confusional State (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Emotional Distress (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0)
Post-Traumatic Stress Disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chronic Kidney Disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Haemoglobinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Micturition Urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oliguria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Renal Failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary Retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Pain (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urine Flow Decreased (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostatic Obstruction (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Testicular Swelling (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 8 (8) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0)
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 0 (0) | 2 (2) | 0 (0)
Paranasal Sinus Discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0)
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Sleep Apnoea Syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillar Inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ingrowing Nail (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Nail Pigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 3 (3) | 0 (0)
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain Of Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Palmar-Plantar Erythrodysaesthesia Syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Precancerous Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2) | 2 (2) | 0 (0)
Pruritus Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash Generalised (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rash Macular (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Seborrhoeic Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin Lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin Mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Swelling Face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Brachiocephalic Vein Thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Flushing (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot Flush (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 5 (5) | 1 (1) | 8 (8) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Systolic Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor supports publication of clinical trial results but may request that investigators temporarily delay or alter publications in order to protect proprietary information. The Sponsor may also require that the results of multicenter studies be published only in their entirety and not as individual site data.

DOCUMENTS (2):
  • Study Protocol (2014-06-16): https://cdn.clinicaltrials.gov/large-docs/40/NCT01587040/Prot_001.pdf
  • Statistical Analysis Plan (2015-07-13): https://cdn.clinicaltrials.gov/large-docs/40/NCT01587040/SAP_000.pdf